CLINICAL TRIAL: NCT01756339
Title: A Randomized, Double-Blind, Multi-Center Study to Evaluate the Efficacy and Safety of Oral Solithromycin (CEM-101) Compared to Oral Moxifloxacin in the Treatment of Adult Patients With Community-Acquired Bacterial Pneumonia
Brief Title: Efficacy and Safety Study of Oral Solithromycin (CEM-101) Compared to Oral Moxifloxacin in Treatment of Patients With Community-Acquired Bacterial Pneumonia
Acronym: SOLITAIRE-ORAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE01-300
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Community-acquired Bacterial Pneumonia
Keywords: Pneumonia; CABP; CAP; Macrolide
MeSH Terms: conditions — Pneumonia | interventions — solithromycin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solithromycin (Experimental): Solithromycin 800 mg orally (PO) on Day 1 followed by 400 mg PO daily on Days 2 through 5, followed by placebo on Days 6 and 7
  Interventions: Drug: Solithromycin; Other: Placebo to match solithromycin
- Moxifloxacin (Active Comparator): Moxifloxacin 400 mg PO daily on Day 1 through Day 7
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Solithromycin
  Other Names: CEM-101
  Arms: Solithromycin
Drug: Moxifloxacin
  Other Names: Avelox
  Arms: Moxifloxacin
Other: Placebo to match solithromycin
  Arms: Solithromycin

SUMMARY:
This study will evaluate the safety and efficacy of an experimental antibiotic, solithromycin, in the treatment of adult patients with community-acquired pneumonia.

DETAILED DESCRIPTION:
Community-acquired bacterial pneumonia (CABP) is an acute infection of the pulmonary parenchyma with symptoms such as fever or hypothermia, chills, rigors, chest pain, and/or dyspnea. The widespread emergence of antibiotic resistant pathogens, including the macrolide-resistant Streptococcus pneumoniae, has resulted in a need for new and effective antibiotics that have activity against CABP pathogens. Solithromycin is a fourth generation macrolide antibiotic with excellent activity against resistant S. pneumoniae and other key typical and atypical bacterial respiratory pathogens. A completed Phase 2 study showed comparable efficacy to levofloxacin in adults with CABP.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age
* An acute onset of at least 3 of the following signs and symptoms (new or worsening):

  1. Cough
  2. Production of purulent sputum
  3. Shortness of breath (dyspnea)
  4. Chest pain due to pneumonia
* At least 1 of the following:

  1. Fever
  2. Hypothermia
  3. Presence of pulmonary rales and/or evidence of pulmonary consolidation
* PORT Risk Class II, III, or IV
* Presence of lobar, multilobar, or patchy parenchymal infiltrate(s) consistent with acute bacterial pneumonia on a pulmonary imaging study
* Not received any systemic antibiotics during the prior 7 days

Exclusion Criteria:

* Ventilator-associated pneumonia
* Known anatomical or pathological bronchial obstruction or a history of bronchiectasis or documented severe chronic obstructive pulmonary disease
* Hospitalization within 90 days or residence in a long-term care facility within 30 days prior to the onset of symptoms
* Presence of known:

  1. Viral or fungal pneumonia
  2. Pneumocystis jiroveci pneumonia
  3. Aspiration pneumonia
  4. Other non-infectious causes of pulmonary infiltrates (e.g. pulmonary embolism, hypersensitivity pneumonia, congestive heart failure)
  5. Primary or metastatic lung cancer
  6. Cystic fibrosis
  7. Active or suspected tuberculosis
* Known HIV or myasthesia gravis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Early clinical response rate in the Intent to Treat (ITT) population | 72 [±12] hours after the first dose of study drug
  To determine noninferiority (NI) in early clinical response rate, in at least 2 of the following 4 cardinal symptoms: cough, shortness of breath, chest pain, and sputum production.

SECONDARY OUTCOMES:
Early clinical response rate in the microITT population | 72 [±12] hours after the first dose of study drug
  To determine NI in early clinical response rate of oral solithromycin compared to oral moxifloxacin in the mITT population
Clinical success rates in the ITT and Clincally Evaluable (CE) populations | 5 to 10 days after the last dose of study drug
  To determine the overall clinical success rates of oral solithromycin compared to moxifloxacin

CONTACTS AND LOCATIONS:
Overall Officials: David Oldach, MD, Study Director — Melinta Therapeutics, Inc.
Locations (87):
- United States (21):
  - Glendale, California
  - Los Angeles, California
  - Mission Hills, California
  - Oxnard, California
  - Pasadena, California
  - Sylmar, California
  - Torrance, California
  - DeBary, Florida
  - DeLand, Florida
  - Miami, Florida
  - Saint Cloud, Florida
  - Tampa, Florida
  - Duluth, Georgia
  - New Bedford, Massachusetts
  - Butte, Montana
  - Columbus, Ohio
  - Downingtown, Pennsylvania
  - Summerville, South Carolina
  - Rapid City, South Dakota
  - Houston, Texas
  - Splendora, Texas
- Argentina (9):
  - La Plata, Buenos Aires
  - Loma Hermosa, Buenos Aires
  - Tandil, Buenos Aires
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
  - Santa Fe, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
  - Buenos Aires
  - Caba
- Bulgaria (4):
  - Pernik, Bulgaria
  - Rousse, Bulgaria
  - Sofia, Bulgaria
  - Sofia
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Cornwall, Ontario
  - Montreal, Quebec
- Beroun, Czechia
- Santo Domingo, Dominican Republic
- Ecuador (3):
  - Guayaquil, Guayas
  - Guayaquil
  - Quito
- Estonia (2):
  - Tallinn
  - Tartu
- Germany (3):
  - Hofheim, De-he
  - Rotenburg (Wümme), De-ni
  - Hanover
- Hungary (3):
  - Budapest
  - Kecskemét
  - Nyíregyháza
- Latvia (3):
  - Daugavpils
  - Liepāja
  - Riga
- Poland (4):
  - Krakow
  - Lodz
  - Lublin
  - Zgierz
- San Juan, Puerto Rico
- Romania (4):
  - Bucharest
  - Craiova
  - Iași
  - Timișoara
- Russia (6):
  - Saint Petersburg, Leningradskaya Oblast'
  - Smolensk, Smolensk Oblast
  - Chelyabinsk
  - Moscow
  - Saint Petersburg
  - Smolensk
- South Africa (12):
  - Thabazimbi, Limpopo
  - Halfway House, Midrand
  - Middelburg, Mpumalanga
  - Witbank, Mpumalanga
  - Korsten, Port Elizabeth
  - Hillcrest, Pretoria
  - Benoni
  - Bloemfontein
  - Cape Town
  - Krugersdorp
  - Pretoria
  - Worcester
- Spain (6):
  - Badalona, Barcelona
  - Majadahonda, Madrid
  - Valencia, Valencia
  - Barcelona
  - Madrid
  - Mataró

REFERENCES:
- [Derived] Barrera CM, Mykietiuk A, Metev H, Nitu MF, Karimjee N, Doreski PA, Mitha I, Tanaseanu CM, Molina JM, Antonovsky Y, Van Rensburg DJ, Rowe BH, Flores-Figueroa J, Rewerska B, Clark K, Keedy K, Sheets A, Scott D, Horwith G, Das AF, Jamieson B, Fernandes P, Oldach D; SOLITAIRE-ORAL Pneumonia Team. Efficacy and safety of oral solithromycin versus oral moxifloxacin for treatment of community-acquired bacterial pneumonia: a global, double-blind, multicentre, randomised, active-controlled, non-inferiority trial (SOLITAIRE-ORAL). Lancet Infect Dis. 2016 Apr;16(4):421-30. doi: 10.1016/S1473-3099(16)00017-7. Epub 2016 Feb 5. PMID 26852726